CLINICAL TRIAL: NCT03321474
Title: Clinical Evaluation of Fracture Resistance and Color Changes of All Ceramic Laminate Veneers Prepared With Modified Gull Wing Versus Conventional Technique
Brief Title: Clinical Evaluation of Fracture Resistance and Color Changes of Laminate Veneer With Gull Wing Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Elshamy, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-10-24
Record Dates: First submitted 2017-10-21; First posted 2017-10-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Discolored Teeth
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified gull wing preparation (Experimental): Gullwing preparation is the inciso - proximal extension of porcelain laminates veneer margin more palatally. The preparation finished at the gingival margin and extended towards the papilla to finish the interproximal elbow preparation
  Interventions: Procedure: modified gull wing preparation
- conventional preparation (Active Comparator): In conventional preparation of veneer it circumvents the contact areas and extends palatally in the incisal third of the tooth only. The preparation thickness is defined by a 0.5 mm facial and 1.5-2.0 mm incisal reduction with the proximal finish lines placed facially to the proximal contacts
  Gull wing (dog leg) preparation is the inciso - proximal extension of porcelain laminates veneer margin more palatally. This preparation design helps to hide the restoration margin when viewed from an angle, especially in discoloration.
  The preparation thickness is defined by a 0.5 mm facial and 1.5-2.0 mm incisal reduction with the proximal finish lines The preparation finished at the gingival margin and extended towards the papilla to finish the interproximal elbow preparation.
  Interventions: Procedure: modified gull wing preparation

INTERVENTIONS:
Procedure: modified gull wing preparation — preparation is the inciso - proximal extension of porcelain laminates veneer margin more palatally.
  The preparation finished at the gingival margin and extended towards the papilla to finish the interproximal elbow preparation.
  Other Names: dog leg ,dog-led -proximal extension preparation

SUMMARY:
Patient with discolored anterior teeth and need conservative restoration treated with all ceramic esthetic laminate veneers. The Patient will be satisfied with restoration mimic the surrounding natural teeth, but conventional preparation shows approximately 60% of veneer failure in form of color change and nearly 67% Fractures of laminate veneers so the modified gull wing preparation is a significant factor affecting the final esthetic especially in discolored teeth and improve fracture resistance of the restoration.

DETAILED DESCRIPTION:
This trial will be conducted on patient from the outpatient clinic in the fixed prosthodontics clinic, faculty of oral and dental medicine, Cairo University Adherence session will take place in the presence of the patients in the initial visit. This include that patient will be informed by Z Elshamy about the study steps and maintenance of oral hygiene instructions. Participants will be asked by Z Elshamy if they have any problems.

Motivation and enforcing the maintenance of oral hygiene measures by ZElshamy.

The visits will be designated as follow:

Visit 1: Preoperative records, face-to-face adherence reminder session, clinical, radiographic examination, intraoral photographs, and primary impression for diagnostic cast construction. Visit 2: teeth preparation, secondary impression using addition silicone rubber base material and temporary restoration. Visit 3: one week after the second visit, try in for the restoration will be done.

Visit 4: placement and permanent cementation of the final restoration. Visit 5: Every 2 months post operatively follow-up visit for one year. Sample size: Since no previously published effect size data regarding the effectiveness of neither the intervention nor the control exist, an estimated sample of (20 restorations) would be used with allocation ratio 1:1 Recruitment: The patients fulfilled the inclusion criteria will be selected from the outpatient clinic of the fixed prosthodontics department - Cairo University. Screening of patients will be carried out until the target population is reached.

Methods: Assignment of interventions (for controlled trial) Sequence generation. The participant teeth will be allocated into two groups with 1:1 allocation ratio by using computerized Sequence generation.

Plans to promote participant retention &complete follow up :

Telephone numbers and address of the patient included in the study will be Recorded. All patients will be given a phone call before the next appointment.

Data management: All data will be entered electronically. Patient files are to be stored in Numerical order in a secured place. This will be carried out by ZElshamy Statistical methods Data analysis All Data will be collected, checked, revised, tabulated and entered into the computer by ZElshamy. Quantitative variables from the normal distribution will be expressed as mean and standard deviation (SD) values. To test the significant differences between two groups at different follow-up period's student t-test will be used. Significant level will be set at P ≤ 0.05 Statistical analysis will be done using Statistical Package for Social Sciences, Version 21.0 (SPSS, IBM, Chicago, III, USA) for Windows. Data monitoring: The main supervisor is responsible for data monitoring if harms arise, an interim analysis will be done. (El Mahallawi O).

Harms: Any adverse effect of pain or even failure will be recorded, documented and treated. Consent: Researcher will discuss the trial with all patients. Patients will then be able to have an informed discussion with the researcher. A researcher will obtain written consent from patients willing to participate in the trial. All consent forms will be in the Arabic language Confidentiality :All study-related information will be stored securely. All participants' information will be stored in locked file cabinets in areas with limited access. All data collection, process, and administrative forms will be identified by a coded ID [identification] number only to maintain participant confidentiality. All records that contain names or other personal identifiers will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems.

Access to data :The investigator and supervisors will be given access to the data sets. All data sets will be password protected. To ensure confidentiality, Participant study information will become confidentially Ancillary and post-trial care :All patients will be followed up until complete period study& patients' satisfactions occur. As any prosthetic treatment post insertion adjustment is necessary and in this trial recalls maintenance.

Dissemination policy : Study results will be published as partial fulfillment of the requirements for PHD degree in fixed prosthodontics.

- Topics suggested for presentation or publication will be circulated to the authors.

Data collection methods:

Primary outcome: The fracture of the restoration of the two groups will be assessed using the modified United States public health service ( USPHS) criteria Secondary outcome: Color changes of the two groups will be assessed using the modified United States public health service (USPHS) criteria

ELIGIBILITY:
* Inclusion Criteria
* age groups from 18-50-year-old
* patients able to read and sign the informed consent.
* patient without periodontal diseases
* Patients indicated for laminate veneers.
* patients Willing to return for follow -up
* Exclusion Criteria
* Patients with poor oral hygiene
* patients with endodontic ally treated teeth
* patients with Psychiatric problems

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
fracture of restoration | one year
  The fracture of the restoration of the two groups will be assessed using the modified United States public health service ( USPHS) criteria

SECONDARY OUTCOMES:
color changed | one year
  Secondary outcome : Color match Color changes of the two groups will be assessed using the modified United States public health service (USPHS) criteria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duzyol M, Duzyol E, Seven N. Fracture Resistance of Laminate Veneers Made with Different Cutting and Preparation Techniques. 2016;4(3):42-48. doi:10.12691/ijdsr-4-3-3.
- [Background] Alhekeir DF, Al-Sarhan RA, Al Mashaan AF. Porcelain laminate veneers: Clinical survey for evaluation of failure. Saudi Dent J. 2014 Apr;26(2):63-7. doi: 10.1016/j.sdentj.2014.02.003. Epub 2014 Mar 26. PMID 25408598